CLINICAL TRIAL: NCT06696560
Title: Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yahia Abd almonem Sayed (Other)
Responsible Party: Sponsor-Investigator, Yahia Abd almonem Sayed, Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries., Assiut University
Organization: Assiut University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AssiutU 1
Record Dates: First submitted 2024-11-12; First posted 2024-11-20 (Actual); Last update posted 2024-11-20 (Actual); Status verified 2024-11

CONDITIONS: Rheumatic Heart Disease With Valvulitis

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries. (Other): Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries.
  Interventions: Other: Minimal Invasive Approaches in Aortic surgeries.

INTERVENTIONS:
Other: Minimal Invasive Approaches in Aortic surgeries. — Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries

SUMMARY:
To compare intraoperative and immediate postoperative outcomes of mini-sternotomy versus mini-thoracotomy as less invasive techniques in patients with isolated aortic valvular and subvalvular disease requiring surgery according to inclusion criteria.

DETAILED DESCRIPTION:
1. It has been demonstrated that minimally invasive aortic valve replacement (MIAVR) approaches are safe and effective for the treatment of aortic valve diseases. To date, the main advantage of these approaches is represented by the reduced surgical trauma, with a subsequent reduced complication rate and faster recovery. This makes such approaches an appealing choice also for frail patients [obese, aged, chronic obstructive pulmonary disease (COPD)(1).
2. Minimally invasive aortic valve replacement (MIAVR) has been increasingly accepted in the surgical community as a potential alternative to conventional sternotomy, with advantages of reduced trauma, improved cosmotic and reduced hospitalization(2).
3. The Mini sternotomy (MS) approach represents the most common technique used for Minimally invasive AVR. The MS approach is achieved through 6 to 10cm midline vertical skin incision, performing a partial J sternotomy at the third to fifth intercostal space (3). MIAVR via right mini thoracotomy (RT) is performed through five to seven cm skin incision placed at the level of the second intercostal space without rib resection. After sacrificing the right internal thoracic artery(4).
4. Despite these excellent results, there have been an increasing number of cases performed via minimally invasive aortic valve replacement (MIAVR). This approach has now become an established alternative to FS in order to reduce the "invasiveness" of the surgical procedure, while maintaining the same efficacy, quality and safety of a conventional approach (5).

ELIGIBILITY:
Inclusion Criteria:

1. Patients with isolated Aortic valve and subvalvular disease.
2. sexes included with acceptance of patients to participate in this study and approval of Ethical Committee.

Exclusion Criteria:

1. Patients ages who less than 16 yrs and more than 60yrs.
2. Emergent open heart surgery.
3. Patients with current Infective endocarditis.
4. Patients with chest deformity pectus excavatum or carinatum due to difficult access.
5. The patient refused to sign the informed consent to participate in the research.
6. Patients with Aortic root abscess or Aortic dilatation at root or ascending parts.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 52 (Estimated)
Dates: Start 2024-11-15 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-01-30 (Estimated)

PRIMARY OUTCOMES:
Minimal Invasive Approaches For Aortic Valvular and Subvalvular Surgeries. | Within 2 years .
  To reduce operation duration,so less hospital stay period. Echocardiography assessment intraoperative and postoperative.